CLINICAL TRIAL: NCT01354769
Title: Capnography Library - Data Collection in the Critical Care Environment Stage 2
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D0006746A
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2011-05

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-intubated patients
  Interventions: Device: CapnoStream20
- Intubated patients
  Interventions: Device: CapnoStream20

INTERVENTIONS:
Device: CapnoStream20 — The monitor used for data gathering is a CapnoStream20-multi parameter monitor
  Other Names: Capnostream Bedside Monitor, Oridion Medical Ltd.

SUMMARY:
Capgnography is the monitoring of the concentration or partial pressure of carbon dioxide in the expired respiratory gases; as such, it is a non-invasive monitoring technique which allows fast and reliable insight into ventilation, circulation and metabolism. Capnography has proven to be more effective than clinical judgement alone in the early detection of adverse respiratory events. The shape of a capnogram is identical in all humans with healthy lungs; any deviations in shape must be investigated to determine a physiological or a pathological cause of the abnormality.

Data from a previous pilot study yielded two major findings:

1. Prediction of requirement for intubation, by the creation of an "Integrated Pulmonary Index" (IPI) based on non-invasive physiological parameters
2. Breathing patterns during weaning in order to identify specific patterns used to predict extubation success/failure

The intent of the current study is to gather sufficient data to either prove or disprove the findings of the previous study

DETAILED DESCRIPTION:
The patient's monitoring period will be as follows:

Non-intubated patients - Initiation: As soon as possible after admission and/or extubation and no later than 24 hours after either. Termination- either 2 hours after intubation or after 8 hours of monitoring overall.

Intubated patients - Initiation: No later than 24 hours after a decision to begin weaning has been made . Termination: Upon ICU (Intensive Care Unit) discharge or for the duration of 10 days at most.

Data will be collected using three tools:

1. CapnoStream raw data (CO2 (Carbon dioxide) waveform, EtCO2 (End-tidal Carbon dioxide), respiratory rate, SpO2 (Saturation of peripheral Oxygen), pulse rate, IPI, alarms, events and any other messages generated by the monitor) will be transferred from the monitor to a laptop via a dedicated recording program.
2. Ventilator data (settings and resultant patient parameters) will be transferred from the monitor to a laptop via a dedicated recording program.
3. Patient monitoring parameters (heart rate, blood pressure, CVP (Central Venous Pressure), temperature, spirometry values etc) shall be recorded from the multi parameter monitors already in use in the ICU and transferred online to a laptop using dedicated recording software.

All recorded parameters will be synchronized. Data will be recorded from at least two of the tools, the Capnostream and the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Suffering from severe illness requiring admission to the ICU
* Expected to be hospitalized in the ICU for a minimum of 8 hours

Exclusion Criteria:

* Under the age of 18
* The patient's refusal to participate in the study
* Any change in the patient's condition that may interfere with data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-intubated and intubated patients being treated for severe illnesses in the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Einav-Bromiker, MD, Principal Investigator — Shaare Zedek Medical Centre
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided